CLINICAL TRIAL: NCT03480698
Title: C-REGS2 - a Registry Study to Observe Clinical Practices, Safety and Efficiency of Routine Use of Cerebrolysin in the Treatment of Patients with Moderate to Severe Neurological Deficits After Acute Ischaemic Stroke
Brief Title: Cerebrolysin REGistry Study in Stroke - a High-quality Observational Study of Comparative Effectiveness
Acronym: C-REGS2
Status: Completed | Type: Observational
Sponsor: Ever Neuro Pharma GmbH (Industry)
Collaborators: IDV Data analysis and study planning Dr. Rahlfs (Unknown)
Responsible Party: Sponsor
Other Study IDs: EVER-AT0717
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — cerebrolysin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cerebrolysin and standard stroke care
  Interventions: Drug: Cerebrolysin
- Standard stroke care

INTERVENTIONS:
Drug: Cerebrolysin — Dosage, frequency, duration and mode of administration of Cerebrolysin follow the local hospital practice in accordance with the terms of the local marketing authorization and is not amended or influenced by the study. Prescribed Cerebrolysin will be used as solution for injection/concentrate for solution for infusion.
  Groups: Cerebrolysin and standard stroke care

SUMMARY:
This study investigates the clinical practices, safety and effectiveness of Cerebrolysin in routine treatment of patients with moderate to severe neurological deficits after acute ischemic stroke.

DETAILED DESCRIPTION:
Patients registered: Acute Ischemic Stroke patients with moderate to severe neurological deficits

All patients receive acute stroke care according to local treatment standards, not amended or influenced by the study:

Cerebrolysin Group:

Patients who are treated with Cerebrolysin; dosage, frequency and duration follows local clinical practice in accordance with terms of the local marketing authorization

Control group:

Patients who are not treated with Cerebrolysin

Observation criteria:

* Signed Informed Consent
* Clinical diagnosis of acute ischemic stroke confirmed by imaging
* Moderate to severe neurological deficits with NIH Stroke Scale (NIHSS) 8 to 15, both inclusive
* No prior stroke
* No prior disability
* Patient's independence prior to stroke onset (pre-morbid mRS of 0 or 1)
* Reasonable expectation of successful follow-up (max. 100 days)

The study follows the recommendations of the Principles for Good Research on Comparative Effectiveness (GRACE).

In order to comply with recent calls for high-quality non-interventional comparative effectiveness research, a risk-based centralized statistical approach to monitoring is introduced in combination with targeted on-site monitoring for ongoing surveillance of study conduct, thus ensuring highest standards of data quality and integrity according to the most recent requirements of the ICH E6 Guideline for Good Clinical Practice (GCP, Amendment R2, July 2015), the FDA Guidance for Industry on a Risk-based Approach to Monitoring, and the EMA reflection-paper on risk-based quality management in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Clinical diagnosis of acute ischemic stroke confirmed by imaging
* Moderate to severe neurological deficits with NIH Stroke Scale (NIHSS) 8 to 15, both inclusive
* No prior stroke
* No prior disability
* Patient's independence prior to stroke onset (pre-morbid mRS of 0 or 1)
* Reasonable expectation of successful follow-up (max. 100 days)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe neurological deficits after acute ischemic stroke (NIHSS 8-15) at baseline
Sampling Method: Non-Probability Sample
Enrollment: 1851 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Ordinal modified Rankin Scale (mRS) at 3 months after stroke onset | 3 months
  The modified Rankin Scale scale is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6, running from perfect health without symptoms to death.

SECONDARY OUTCOMES:
Ordinal NIH Stroke Scale (NIHSS) at 21 days and 3 months after stroke onset | Day 21 and 3 months
  The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Ordinal modified Rankin Scale (mRS) at 21 days after stroke onset | 21 days
  The modified Rankin Scale scale is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6, running from perfect health without symptoms to death.
Proportion of patients with excellent recovery (mRS score 0-1) at 3 months after stroke onset | 3 months
  The modified Rankin Scale scale is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6, running from perfect health without symptoms to death.
Proportion of patients with functional independence (mRS score 0-2) at 3 months after stroke onset | 3 months
  The modified Rankin Scale scale is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6, running from perfect health without symptoms to death.
Ordinal MoCA at 3 months after stroke | 3 months
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. The MoCA test is a one-page 30-point test administered in approximately 10 minutes. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brainin, Univ.-Prof. Dr., Study Director — Danube University Krems - Head of the Department for Clinical Neuroscience and Preventive Medicine / Head of the Center for Neurosciences
Locations (8):
- Austria (8):
  - Landesklinikum Amstetten, Amstetten
  - Krankenhaus der Barmherzigen Brüder Eisenstadt, Eisenstadt
  - Universitätsklinik Innsbruck, Innsbruck
  - Kepler Universitätsklinikum, Linz
  - CDK Salzburg, Universitätsklinik für Neurologie, Salzburg
  - UK St. Pölten, Sankt Pölten
  - UK Tulln, Tulln
  - LK Wiener Neustadt, Wiener Neustadt

IPD SHARING:
Plan to Share IPD: No